CLINICAL TRIAL: NCT01865045
Title: Pharmacogenetics of Vinorelbine in Malignant Pleural Mesothelioma Patient
Brief Title: Pharmacogenetics Of Vinorelbine In Malignant Pleural Mesothelioma Patients
Status: Completed | Type: Observational
Sponsor: Armando Santoro, MD (Other)
Responsible Party: Sponsor-Investigator, Armando Santoro, MD, Principal Investigator, Istituto Clinico Humanitas
Organization: Istituto Clinico Humanitas (Other)
Other Study IDs: ONC/OSS-02/2012
Record Dates: First submitted 2013-05-27; First posted 2013-05-30 (Estimated); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Malignant Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no treatment: no treatment

SUMMARY:
This is a multicenter retrospective analysis .The aim of the present study is to investigate the molecular predictors of vinorelbine response in tumor samples of a series of MPM patients and evaluate the possible impact on clinical outcome.

Sample size: around 150 patients based on the availability of tumor size

DETAILED DESCRIPTION:
Vinorelbine has recently become an alternative option for palliation in selected pemetrexed-pretreated patients with malignant pleural mesothelioma (MPM). However, nowadays there are no definitive data about vinorelbine predictors of response in MPM patients. The identification of molecular predictors of effective therapy is important for maximizing therapeutic efficacy and minimizing useless treatment in cancer patients.

In oncology a pharmacogenetic approach to customize the chemotherapy treatment according to individual as well as tumour genetic characteristics represents a modern and intriguing challenge. Recent studies have suggested that the expression levels of class III β-tubulin (TUBB3) or BRCA1, are related to a survival benefit from vinorelbine chemotherapy among patients with advanced solid malignancies, especially non-small cell lung cancer. There are no data about the predictive factors to vinorelbine in MPM patients. The identification of molecular predictors of effective therapy may allow in the future the development of better therapies.

ELIGIBILITY:
Inclusion Criteria:

* MPM patients treated with vinorelbine in the ≥ second line setting will be retrospectively analyzed
* Patients will be selected based on the availability of tumor tissue

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Malignant pleural mesothelioma patients treated with vinorelbine as a second or later line chemotherapy with at least an objective response evaluation.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-11; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Expression of TUBB3 and BRCA1 in MPM tumor tissue by immunohistochemistry and RT-PCR. | 2 months

SECONDARY OUTCOMES:
Association of expression of TUBB3 and BRCA1 with clinical outcome (response, survival) . | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: armando santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
not planned